CLINICAL TRIAL: NCT06898034
Title: Postpartum Ultrasound Evaluation to Assess Risk of Hemorrhage
Status: Recruiting | Type: Observational
Sponsor: Endeavor Health (Other)
Responsible Party: Principal Investigator, Emmet Hirsch, Principal Investigator, Endeavor Health
Other Study IDs: STUDY00000080
Record Dates: First submitted 2025-03-07; First posted 2025-03-27 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Pregnancy Related; Post Partum Hemorrhage
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Ultrasound — Postpartum ultrasound exam

SUMMARY:
Up to 5% of patients in the United States have a postpartum hemorrhage. "Postpartum hemorrhage" means excessive bleeding after delivery. The majority of these bleeds occur immediately with delivery.

The current study focuses on hemorrhages that occur in the "medium-term" (1.5-24 hours after delivery). Investigators are examining whether ultrasound exams performed at the beginning of this period 1.5 to 2 hours after birth can identify markers that predict a medium-term bleed. Data collected for this study will include medical and obstetrical history, details about the course and outcomes of patients' labor and delivery, and particulars about postpartum bleeding. This information will be collected through the end of the patients' delivery admission and will allow correlation with the results of the ultrasound exam. If patients are re-admitted to the hospital after the delivery discharge, investigators may also collect relevant information about those admissions up to 6 weeks postpartum.

All patients after term delivery (≥ 37 weeks' gestation) will be eligible to participate. Patients will be approached to provide consent for participation as early as feasible during a prenatal visit (≥ 36 weeks' gestation) or during the delivery admission. No subjects will be consented while in significant pain, >6cm dilated without an epidural, or >8cm dilatated with an epidural.

ELIGIBILITY:
Inclusion Criteria:

* Currently pregnant and planning to deliver at Endeavor Health >37 weeks gestational age
* English speaking
* Labor <6cm dilated at time of consent without epidural
* Labor <8cm dilated at time of consent with epidural

Exclusion Criteria:

* Preterm delivery
* Non-English speaking
* Any conditions that impairs potential participants decision making

Min Age: 17 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All patients admitted to Labor and Delivery for term delivery at Evanston, Highland Park or Swedish Hospitals (≥ 37 weeks' gestation at any maternal age, not decisionally impaired) will be eligible to participate.
Sampling Method: Non-Probability Sample
Enrollment: 1725 (Estimated)
Dates: Start 2025-03-10 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Ultrasound exam: uterine measurements | From enrollment to 1.5-2 hours post partum
  * Uterine length (cm)
  * Uterine width (cm)
  * Uterine height (cm)
  These will be correlated with subsequent clinical outcomes, including bleeding events.
Ultrasound exam: endometrial stripe | From enrollment to 1.5-2 hours post partum
  Width (cm) of the endometrial stripe (measuring displacement of the uterine walls by intrauterine contents (blood, clots, retained placental fragments or other) to include Doppler study) at 3 levels:
  * Fundal
  * Lower uterine segment
  * Cervix
  These will be correlated with subsequent clinical outcomes, including bleeding events.
Ultrasound exam:fibroids | From enrollment to 1.5-2 hours post partum
  Presence of uterine fibroids (number and size in cm of each)
  These will be correlated with subsequent clinical outcomes, including bleeding events.
Ultrasound exam: Vagina | From enrollment to 1.5-2 hours post partum
  Caliber of the vagina (cm) (to assess distension by clot)
  These will be correlated with subsequent clinical outcomes, including bleeding events.
Ultrasound exam: Bladder | From enrollment to 1.5-2 hours post partum
  * Bladder length (cm)
  * Bladder height (cm)
  * Bladder width (cm)
  All other aspects of clinical management will be left to the discretion of the clinical team.
  These will be correlated with subsequent clinical outcomes, including bleeding events.

SECONDARY OUTCOMES:
Chart review | From enrollment to 6 weeks post partum
  Outcome measures for this study will include details about the postpartum course up to 6 weeks postpartum. This will allow correlation with the results of the ultrasound exam. If patients are re-admitted to the hospital after the delivery discharge, investigators will also collect relevant information about those admissions.

CONTACTS AND LOCATIONS:
Locations (1):
- Endeavor Health, Evanston, Illinois, United States

IPD SHARING:
Plan to Share IPD: No